CLINICAL TRIAL: NCT05485714
Title: Non-invasive Prediction of Esophageal Varices in Patients With Non-Alcoholic Fatty Liver Disease With Advanced Fibrosis; A Single Centre United Arab Emirates Experience
Brief Title: Non-invasive Prediction of Esophageal Varices in Patients With Non-Alcoholic Fatty Liver Disease With Advanced Fibrosis
Status: Completed | Type: Observational
Sponsor: United Arab Emirates University (Other)
Collaborators: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Other Study IDs: UAEU_TWM_MF2058-2022-856
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Varices; Non-alcoholic Fatty Liver; Compensated Cirrhosis
Keywords: Platelet count; Spleen diameter; Baveno VI; non-invasive prediction; liver Stiffness; varices needing treatment; Endoscopy
MeSH Terms: conditions — Esophageal and Gastric Varices; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with non-alcoholic fatty liver with advanced liver fibrosis: Patient with non-alcoholic fatty liver with advanced liver fibrosis with F3 or F4 stage on Fibroscan without any evidence of previous decompensation like ascites, jaundice or encephalopathy
  Interventions: Other: Reviewing records retrospectively of patients undergoing screening endoscopy

INTERVENTIONS:
Other: Reviewing records retrospectively of patients undergoing screening endoscopy — Reviewing records retrospectively of patients undergoing screening endoscopy to assess Baveno VI, expanded Baveno VI, Platelet count/spleen diameter and other non-invasive predictors of esophageal varices or varices needing treatment

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is defined as accumulation of fat in the liver which is not related to either alcohol excess or other causes such viral infection, immune-mediated, or medication related which can lead to fibrosis and later-on, cirrhosis. Over the last years NAFLD related liver cirrhosis has become the commonest cause of chronic liver disease worldwide. Portal hypertension is the major complication caused by increased splanchnic blood flow which leads to development of oesophageal varices (OV). Almost all of the patients with portal hypertension can develop OV sometime in their life and one third of those will bleed, hence identifying the presence of OV is a an important aspect of diagnostic workup of these patients with portal hypertension.

Upper digestive camera test/endoscopy is the only means to diagnose and grade OV but endoscopy is an invasive procedure and its cost effectiveness for screening is also questionable. These limitations and the ever-increasing workload on endoscopy units has led many researchers to identify some parameters that can non-invasively diagnose OV. Researchers have proposed use of platelet count/spleen diameter ratio, liver stiffness on Fibroscan among many non-invasive tools to predict OV in patients with portal hypertension with success. Recently criteria proposed in Baveno VI conference, (Baveno-IV Criteria) recommended that screening endoscopy can be avoided in patients with compensated advanced chronic liver disease (cACLD) with liver stiffness measurement (LSM) less than 20 kPa and a platelet count more than than 150,000/μL with an expanded Baveno-IV criteria suggesting platelet count >110 × 109 cells/L and LSM <25 kPa can spare even more endoscopies with a risk of missing varices needing treatment (VNT) being minimal.

DETAILED DESCRIPTION:
Background:

Non-alcoholic fatty liver disease (NAFLD) is defined as fatty infiltration of the liver not related to alcohol excess or other usual causes of hepatic steatosis e.g. viral or autoimmune hepatitis or secondary to medications and includes a spectrum ranging from steatosis, steatohepatitis, and fibrosis to cirrhosis; and is now the most common cause of chronic liver disease worldwide with prevalence of up to 30%. Although most patients with NAFLD may not progress to advanced fibrosis or cirrhosis, but as it has become so prevalent that still many patients develop cirrhosis and is now a leading indication for liver transplantation in Europe. In terms of global prevalence of NAFLD, it is quite high (32%) in the Middle East region. Portal hypertension is the major complication caused by increased splanchnic blood flow secondary to vasodilation and increased resistance to blood flow through periportal fibrosis which leads to development of oesophageal varices (OV). An estimated 90% of the portal hypertension patients will develop OV sometime in their life and 30% of those will bleed. Moreover 5-50% of the patients with acute variceal bleed will die within first days of the initial episode,6 hence identifying the presence of OV is a fundamental part of diagnostic workup of portal hypertension patients.

Upper digestive endoscopy is the only means to diagnose and grade OV but endoscopy is an invasive procedure and its cost effectiveness for screening is also questionable. These limitations and the ever-increasing workload on endoscopy units has led many researchers to identify some parameters that can non-invasively diagnose OV. The factor most commonly associated with varices in most of these studies was thrombocytopenia, though it lacked sensitivity and specificity. Previously researchers proposed normalizing the platelet count to ultrasonographic spleen diameter and used platelet count/spleen diameter ratio of 909 to predict OV non-invasively in patients with portal hypertension, with 100% prevalence adjusted negative predictive value, and further validation studies showed the generalisability of results. Recent criteria in Baveno-IV conference, (Baveno-IV Criteria), recommends that screening endoscopy can be avoided in patients with compensated advanced chronic liver disease (cACLD) with liver stiffness measurement (LSM) less than 20 kPa and a platelet count more than than 150,000/μL. A new expanded Baveno-IV criteria suggesting platelet count >110 × 109 cells/L and LSM <25 kPa, likely to spare even more endoscopies with a risk of missing varices needing treatment (VNT) of only 1.6% (95% confidence interval, 0.7%-3.5%) in patients within the criteria and 0.6% (95% confidence interval, 0.3%-1.4%) in the overall population of 925 patients with cACLD.

Aim:

The purpose of this study is to compare the ability of various non-invasive methods including Baveno-IV & expanded Baveno-IV criteria, platelet count/spleen diameter, and platelet count/(spleen diameter + LSM), in prediction of VNT in NAFLD with advance liver fibrosis

Patients & Methods:

We plan to include minimum 100 patients of NAFLD related liver fibrosis as per selection criteria

All the patients with NAFLD related liver fibrosis confirmed on Fibroscan referred to Endoscopy Unit, Tawam Hospital for screening of esophageal varices fulfilling the selection criteria will be selected from medical records and their documented demographic data and data pertaining to history of present illness and positive physical signs will be obtained. The biochemical workup (bilirubin, prothrombin time, albumin, creatinine), ultrasound for presence of ascites and bipolar splenic diameter, and data for liver stiffness measurement and results of upper GI endoscopy will be obtained. The Baveno-IV criteria and expanded Baveno-IV criteria and platelet count (in /mm3) to spleen diameter (in mm) ratio will be calculated/applied in all these patients and compared with outcomes of gold standard i.e Endoscopy results. All this information will be collected in excel sheet for further transfer on statistical software for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed to have non-alcohol fatty liver disease
* Evidence of Liver stiffness measurement of > 9.9 KPa (indicative of >F3 fibrosis ).
* Periportal hepatic fibrosis and liver echotexture changes confirmed by an experienced radiologist with expertise in Ultrasound.
* Vitally stable patients (without massive bleeding, encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome, shock).
* Compensated Liver cirrhosis (no evidence of decompensation previously)

Exclusion Criteria:

* Active alcohol abuse (abstinence of alcohol for less than six months).
* Evidence of other etiology for liver cirrhosis like viral infection (HBsAg +ve or Anti-HCV seropositivity or viral DNA seen in past/present) or immune/ congenital cause of liver cirrhosis (like autoimmune, congenital hepatic fibrosis etc)
* Co-morbid liver or biliary disease (hepatoma, biliary channel obstruction).
* Evidence of band ligation/sclerotherapy, portosystemic shunting procedure or surgery for portal hypertension in the past

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with Non-alcoholic fatty liver related advanced liver fibrosis confirmed on Fibroscan (stage F3 or F4) referred to Endoscopy Unit Tawam Hospital, Al Ain Abu Dhabi for screening of esophageal varices fulfilling the above-mentioned criteria will be selected. All consecutive patients over the last five years will be selected
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Comparing non-invasive parameters with gold standard Endoscopy in prediction of esophageal varices in patients with fatty liver with advanced fibrosis | Chart review of selected patients who underwent screening endoscopy over the last 5 years; to be completed in 6 months
  To compare various previous known non-invasive predictors of esophageal varices and compare their ability to predict esophageal varices when compared to gold standard i.e. endoscopy.
  The predictors include;
  1. Platelet count to ultrasonographic spleen diameter ratio ((N/mm3)/mm) of > 909 suggesting esophageal varices are unlikely
  2. Baveno VI criteria i.e. liver stiffness measurement (LSM) less than 20 kPa and a platelet count more than than 150,000/μL suggesting esophageal varices are unlikely 3 New expanded Baveno VI criteria i.e. platelet count >110 × 109 cells/L and LSM <25 kPa suggesting esophageal varices are unlikely

SECONDARY OUTCOMES:
Assessing a new non-invasive parameters with gold standard Endoscopy in prediction of esophageal varices in patients with fatty liver with advanced fibrosis | 6 months
  To look at various previous suggested predictors and see if there is cut off that exists for a new predictor that involves that all three know risk factors for esophageal varices i.e. Platelet count, spleen diameter on ultrasound and liver stiffness in kPa on fibroscan in the form of novel platelet count/(spleen diameter and Liver stiffness measurement) [(N/cm3)/(cm +kpa)] and compare with with gold standard Upper GI Endoscopy to see if this tool can predict the absence of varices needing treatment in patient with fatty liver and advanced hepatic fibrosis (fibrosis stage F3 or F4) in a tertiary care hospital in Al Ain, Abu Dhabi, United Arab Emirates.

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

REFERENCES:
- [Background] Agha A, Anwar E, Bashir K, Savarino V, Giannini EG. External validation of the platelet count/spleen diameter ratio for the diagnosis of esophageal varices in hepatitis C virus-related cirrhosis. Dig Dis Sci. 2009 Mar;54(3):654-60. doi: 10.1007/s10620-008-0367-y. Epub 2008 Jul 2. PMID 18594972
- [Background] Agha A, Abdulhadi MM, Marenco S, Bella A, Alsaudi D, El-Haddad A, Inferrera S, Savarino V, Giannini EG. Use of the platelet count/spleen diameter ratio for the noninvasive diagnosis of esophageal varices in patients with schistosomiasis. Saudi J Gastroenterol. 2011 Sep-Oct;17(5):307-11. doi: 10.4103/1319-3767.84483. PMID 21912056
- [Background] Giannini E, Botta F, Borro P, Risso D, Romagnoli P, Fasoli A, Mele MR, Testa E, Mansi C, Savarino V, Testa R. Platelet count/spleen diameter ratio: proposal and validation of a non-invasive parameter to predict the presence of oesophageal varices in patients with liver cirrhosis. Gut. 2003 Aug;52(8):1200-5. doi: 10.1136/gut.52.8.1200. PMID 12865282
- [Background] Pizzamiglio M, Weicker A, de Terwangne C, Henrion J, Descamps OS, De Vos M. Validation of Baveno VI and Expanded-Baveno VI Criteria for predicting gastroesophageal varices in patients with alcoholic and non-alcoholic fatty liver disease. Acta Gastroenterol Belg. 2022 Apr-Jun;85(2):321-329. doi: 10.51821/88.2.9553. PMID 35709776